CLINICAL TRIAL: NCT02402335
Title: Study of Different Types of Pains in Groups of Patients With Different Diagnoses of Degenerative Diseases and Their Related Surgeries
Brief Title: Study of Different Types of Backache in Groups of Patients With Different Diagnoses of Degenerative Diseases
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Bonn (Other)
Responsible Party: Principal Investigator, Robert Pflugmacher, PD Dr med Robert Pflugmacher, University Hospital, Bonn
Other Study IDs: UKBORTAB01
Record Dates: First submitted 2015-03-18; First posted 2015-03-30 (Estimated); Last update posted 2015-03-30 (Estimated); Status verified 2015-03

CONDITIONS: Ache
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1 Fracture of vertebra: Osteoporotic fracture of the vertebra
- 2 Nerve Compression: Osteochondria, Spinal disc herniation, Nerve compression

SUMMARY:
The purpose of this study is to examine whether there are relations between different types of pain in groups of patients with different diagnoses of degenerative diseases of the spinal column and their related surgeries.

DETAILED DESCRIPTION:
In the context of this work the pain of different groups of patients should be examined by means of the painDetect Questionnaire, the Roland-Morris disability questionnaire, clinical examinations and different imaging procedures. Two groups of patients are compared with each other. Group one consists of patients with osteoporotic fractures of the vertebra. Group two is formed by patients with osteochondria , spinal disc herniation and nerval compression. Both groups of patients undergo surgery, as they are suffering from pain (e.g. kyphoplasty, nucleotomy, spondylodesis, decompression). In order to differentiate between chronic nociceptive pain and chronic neuropathic pain in these two groups the painDetect questionnaire is used. To examine the severity of disability in the patients' everyday life the Roland-Morris Disability questionnaire is used.

The included patients are examined and seen preoperative, postoperative before discharge from hospital, 6 weeks and 6 months after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Backache because of degenerative diseases
* Surgery is necessary

Exclusion Criteria:

-

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients of the University Hospital of Bonn who are strongly suffering from backaches that cannot be treated anymore by conservative methods.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2015-02; Primary Completion 2016-10 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Backache objectified by the PainDETECT Questionnaire | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Robert Pflugmacher, PD Dr med, Principal Investigator — University Hospital Bonn, Clinics of Orthopedics and Traumatology
Locations (1):
- University Hospital of Bonn, Bonn, North Rhine-Westphalia, Germany